CLINICAL TRIAL: NCT04778462
Title: Effect of High- Power Pain Threshold Ultrasound Versus Extracorporeal Shock Wave on Myoelectric Activity of Upper Trapezius Myofascial Trigger Point
Brief Title: Myoelectric Activity of Upper Trapezius Trigger Point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Hager Mahomud Mohamed elsayed, Principle investigator, MTI University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Mti
Record Dates: First submitted 2021-02-18; First posted 2021-03-03 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Trigger Point Pain, Myofascial
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: 1. sixty subjects from both genders with their age between 20 and 26 years old
  2. Symptoms of active TrPs unilateral on at least one side of the upper fiber of trapezius muscle presence of at least one trigger point symptoms lasting from 0 to 2 weeks age
  3. The patients will be randomly assigned into three different groups Group (A) will receive extracorporeal shock wave plus stretch, strength exercise and ischemic compression Group (B) will receive high-power pain threshold ultrasound plus stretch, strength exercise and ischemic compression Group (C) will receive conventional treatment (stretch, strength exercise and ischemic compression.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extracorporeal shock wave (Experimental): Extracorporeal shock wave group A consist of 15 subject will receive extracorporeal shock wave and conventional treatment for trigger points for two weeks four treatment sessions
  Interventions: Device: extracorporeal shock wave and conventional treament
- High-power pain thershold ultrasound (Experimental): High -power pain thershold group b consist of 15 subject will receive high power pain threshold ultrasound and conventional treatment for upper trapezius trigger points for two weeks four treatment session
  Interventions: Device: high pain threshold ultrasound and conventional treatment for myofascial pain syndrome trigger points
- Controlled group (Other): controlled group consist of 15 subjects will receive conventional treatment for trigger point for two weeks
  Interventions: Other: conventional treatment for myofascial pain trigger point

INTERVENTIONS:
Device: extracorporeal shock wave and conventional treament — Extracorporeal shock wave for 700 impulses of 0.056 mJ/mm at a frequency of 10 Hz to the taut band and 300 impulses surrounding the taut band will be applied as low energy 2 sessions per week for 2 weeks The will be used as a radial type of shock wave therapy.
  Strengthening, stretching exercises and ischemic compression:
  1. Isometric neck extensor exercise:
  2. Isometric neck flexor exercise:
  3. Isometric neck side bending muscle exercise:
  Stretching exercise:
  Passive stretching for the neck extensor muscles:
  Passive stretching of the neck side-bending muscles:
  Ischemic compression
  Other Names: extracorporeal shock wave
  Arms: Extracorporeal shock wave
Device: high pain threshold ultrasound and conventional treatment for myofascial pain syndrome trigger points — will be applied in continuous mode, with the probe placed directly on the TrP and held motionless. To elicit threshold pain, the US probe will be kept static on the TrP. Intensity gradually will be increased to the level of maximum pain the patient could bear. It will be kept at that level for 3 to 4 seconds, then will be reduced to the half-intensity level for another 15 seconds. This procedure was repeated 3 times.the intensity of US will be dependent on the patient's level of pain. intensity will be applied in the range of 0.5 to 2.0 Watt per/cm2. Patients continually report their pain level and its localization and nature High-power pain threshold US will be applied 4 times, with a 3-day interval 2 sessions per week for 2 weeks .
  1)Isometric neck extensor exercise2)Isometric neck flexor exercise3)Isometric neck side bending muscle exercise,Stretching exercise:Passive stretching for the neck extensor muscles ,stretching of the neck side-bending muscles,Ischemic compression
  Other Names: HPPT
  Arms: High-power pain thershold ultrasound
Other: conventional treatment for myofascial pain trigger point — Strengthening, stretching exercises and ischemic compression:
  1. Isometric neck extensor exercise:
  2. Isometric neck flexor exercise:
  3. Isometric neck side bending muscle exercise:
  Stretching exercise:
  Passive stretching for the neck extensor muscles:
  Passive stretching of the neck side-bending muscles:
  Ischemic compression
  Arms: Controlled group

SUMMARY:
Myofascial trigger points are a muscular dysfunction at the level of the motor end-plate and the sarcoplasmic reticula that, in turn, cause a local contraction with ischemia -induced hypoxia. Along with the hypoxia, the resulting energy crisis leads to a sensation of the surrounding nociceptors . Extracorporeal shock wave therapy (ESWT) is recently considered an effective treatment for myofascial pain syndrome. It's been proved an effective in musculoskeletal disease fasciitis

. It is significant since it is a non-invasive and simple treatment, easy to apply at a large surface, and has fewer side effects with low intensity even if it requires relatively high cost, ESWT has been proved to be more effective than conventional ultrasound on MTrPs in the upper trapezius muscle and showed that ESWT is more effective

. It has been found that three sessions of ESWT significantly improved pain levels, neck disabilities, and the quality of life by reducing the number of MTrPs .

ESWT could reduce the pain of myofascial pain syndrome by pain signal alteration, promoting angiogenesis and increasing perfusion in ischemic tissues induced by sensitization of nociceptors and muscle ischemia.

Ultrasound with deep heat is used in treatment of myofascial trigger point due to the properties of achieving vasodilation, accelerating the metabolism, increasing viscoelasticity and reducing pain and muscle spasm

High power pain threshold ultrasound found to be effective in many literatures in treatment of myofascial trigger point

. Study was performed comparing effect of high power pain threshold ultrasound with conventional ultrasound proved that high power pain threshold is more effective in treating upper trapezius myofascial It was found in the treatment of MPS, HPPT US therapy could be considered as a reliable and more effective and has positive effect method than low-dose and conventional US therapies

This study will be presented as a part of ongoing study. The ongoing study investigates the effect of different intensities of ultrasound on upper trapezius trigger points. The current study will investigate the myoelectric activities of trigger points after application of high power pain threshold ultrasound

DETAILED DESCRIPTION:
Myofascial pain is defined as pain that originates from myofascial trigger points in skeletal muscle. It is prevalent in regional musculoskeletal pain syndromes, either alone or in combination with other pain generators Myofascial pain syndrome is represented by many clinical symptoms such as pain, hyperirritable nodule of spot tenderness, referred pain, and muscle spasm by trigger points. The upper trapezius is probably the muscle most often beset by trigger points It was assumed that the muscle fibers are shortened and taut bands are made by calcium influx in damaged fibers or acetylcholine secretion in motor end plates. The trigger points are the hyperirritable nodules of spot tenderness in a palpable taut band of skeletal muscle that may cause pain to a distant point and also causes distant motor and autonomic effects Once myofascial trigger points are activated, changes in the structural characteristics and contraction function of the muscle will occur. The most distinctive changes are taut bands, tender nodules, referred pain, local twitch response, muscle weakness, and restricted range of motion Patients with unilateral pain of an upper trapezius muscle exposed to a fatiguing load analyzed with surface electromyography (sEMG) were found to have a difference in sEMG response between healthy and symptomatic muscle Surface electromyography (EMG) analyzes functional changes in muscle by measuring quantitative changes in motor unit action potential that is activated by muscle contraction

Surface EMG, which was used to evaluate the functionality of trigger points in this study, is nonintrusive and convenient; thus, it is widely used in studies on the functional characteristics of muscle, by analyzing the electrical activity of muscle Surface EMG recording fortrigger points shows changes in recruitment of fast-twitch muscle fibers and conduction velocity of motor unit action potential According to Gemmell and Bagust (2009) EMG recordings confirm increased spontaneous activity of motor units in patients with myofascial pain during the "resting state" of muscles.

The treatments of myofascial pain are divided into the invasive and the non-invasive therapy. The invasive therapy is about the injection of medications, dry needling and non-invasive therapy refers to massage, stretching and ultrasound Extracorporeal shock wave therapy (ESWT) is recently considered an effective treatment for myofascial pain

, It is a non-invasive and simple treatment, easy to apply at a large surface, and has fewer side effects with low intensity even if it requires relatively high cost.

ESWT could reduce the pain of myofascial pain syndrome by pain signal alteration, promoting angiogenesis and increasing perfusion in ischemic tissues induced by sensitization of nociceptors and muscle ischemia .

High power pain threshold ultrasound resolve acute active trigger points . High power-pain threshold ultrasound efficient method for relieving painand disability and increasing range of motion Although signiﬁcant in decreasing tissue stiffness Previous study, which is the ﬁrst to make a combined evaluation of the effectiveness of low-, moderate- and high dose (HPPT) US therapies in MPS, the results obtained considered signiﬁcantly in that greater improvements in clinical parameters were generally determined going from low dose to high dose and that the effect was achieved in only four sessions of HPPT US therapy. the cycle of pain-spasm-ischemia-pain is more effectively resolved when the dosage of US, applied for the treatment of trigger points in MPS, is increased the cycle of pain-spasm-ischemia-pain is more effectively resolved when the dosage of US, applied for the treatment of trigger points in MPS, is increased. Therefore, HPPT US therapy can be considered as a more economical treatment than conventional US treatments due to less number of treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

* Both genders will be included with their age between

  . •Symptoms of active TrPs unilateral on at least one side of the upper fiber of trapezius muscle presence of at least one trigger point symptoms lasting from 0 to 2 weeks age
* Subjects have pain at rest, local twitch response, jump sign, limited range of motion and referred pain lies over the lateral aspect of the upper trapezius fiber and superiorly to the ipsilateral occiput .

Exclusion Criteria:

Exclusion Criteria:

* patients who had medication or other therapies for myofascial pain syndrome (Ji Hm et al., 2012) (2)
* patients who had neurological deficits involving the upper limbs, advance osteopathic or arthropathic disorders of the cervical spine or the shoulder of the investigated side
* contraindication of ESWT such as hypertension, coagulopathy, ulcer, recent severe hemorrhage, neoplasm, renal insufficiency, severe hepatic disease, epilepsy, cutaneous pathology, central pain, pregnancy and mental retardation
* The presence of previously diagnosed disease such as (diabetes mellitus, fibromyalgia, hormonal disorder hypothyroidism, hyperthyroidism and rheumatoid arthritis

Ages: 20 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
surface electromyography | before treatment and after 2 weeks of treatment
  change in electrical activity of Trigger points of upper trapezius using surface electromyography
pressure algometer | before treatment and 2 weeks after treatment
  change in pressure pain threshold for upper trapezius trigger
Neck disability index | before treatment and 2 weeks after treatment
  change in the neck function scale contain 10 category each category contains six choices from zero to five ,score from zero to four no disability from five to fifteen this is mild,from fifteen to twenty-four this is moderate, from twenty-five to thirty-four this is severe

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy modern University for technology and science, Cairo, Egypt